CLINICAL TRIAL: NCT01484509
Title: The Estimation of Ambulation Capacity by History Questionnaire (EACH-Q): An Assessment of Its Validity and Inter-day Reproducibility in Patients With Vascular-type Claudication
Brief Title: Subjective and Objective Methods of Assessing Walking Limitation Due to Claudication
Status: Completed | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Sheffield Hallam University (Other); University Hospital, Angers (Other Government); Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: STH16036
Record Dates: First submitted 2011-11-24; First posted 2011-12-02 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2011-11

CONDITIONS: Intermittent Claudication
Keywords: walking impairment; claudication; treadmill; questionnaire
MeSH Terms: conditions — Intermittent Claudication

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Intermittent claudication

SUMMARY:
Leg artery disease is a common condition in which fatty deposits develop in the blood vessels that supply the legs. Many patients with leg artery disease experience a cramp-like leg pain during walking that is relieved by rest; this is called intermittent claudication. To help determine the severity of leg artery disease, patients may be questioned about how far they can walk before claudication pain forces them to stop. However, this information is usually of limited use because most patients poorly estimate their walking capacity. The investigators have developed a simple questionnaire to help estimate walking capacity in patients with leg artery disease. The purpose of this study is to test the validity and reliability of this questionnaire. By validity, the investigators mean the extent to which the questionnaire measures what it is supposed to measure (walking capacity). By reliability, the investigators mean the extent to which the questionnaire produces the same results over time when completed on two different days.

The investigators hypothesise that the investigators simple questionnaire will be valid and reliable.

DETAILED DESCRIPTION:
Claudication is a chronic condition that impairs walking capacity. Lower-extremity peripheral arterial disease (PAD) is a frequent cause of claudication. Claudication is suspected to be vascular-type (i.e. of arterial origin) when pain or discomfort occurs in the leg muscles during exercise and is relieved within 10 min of rest. The "maximal walking distance" (MWD; the distance at which pain forces the patient to stop walking) is of great importance for assessing the severity of claudication. Patient interview is the most readily accessible way of estimating walking capacity in routine clinical practice; however, patients with PAD typically poorly estimate their walking capacity. Open questions about the distance a patient can walk before limb pain or discomfort forces them to stop lack standardisation. Questions such as "Because of a health or physical problem, do you have any difficulty walking for one mile?" only allow for a yes/no response. The functional status component of the 86-item PAVK-86 questionnaire appears useful for estimating MWD, but this is a time-consuming tool. The Walking Impairment Questionnaire (WIQ), which was proposed over a decade ago to standardise the estimation of walking capacity by patient interview, is widely used. However, the WIQ is also relatively complex (14 items with 5 possible answers for each item: 70 boxes), which often results in a large number of errors when self-completed by the patient. Furthermore, the WIQ score is difficult to obtain by mental calculation.

The investigators have developed a simple, 4-item questionnaire, called the Estimation of Ambulation Capacity by History Questionnaire (EACH-Q), for estimating walking capacity in patients with symptomatic PAD (vascular-type claudication). The EACH-Q estimates the maximal duration that can be achieved (8 possibilities ranging impossible to 3 hours or more) at 4 different displacement speeds (from slow walking to running). Scores can be obtained easily by multiplying the rank of each possible answer (impossible being zero) by a speed factor. We recently validated the EACH-Q against constant-load treadmill-walking-test performance in patients suffering from vascular-type claudication. However, further research is needed to assess the validity of the EACH-Q against other objective tests of walking capacity (e.g. incremental treadmill-walking test, 6-min walk test), and to assess its reproducibility.

Hence, the aims of this study are: (i) to assess the validity of the EACH-Q against objective measures of walking capacity obtained from the Gardner-Skinner incremental treadmill-walking test and the 6-min walk test, and; (ii) to assess the inter-day reproducibility of the EACH-Q. The results will be compared against those obtained from the WIQ, and the participant cohort will be patients suffering from vascular-type claudication.

ELIGIBILITY:
Inclusion Criteria:

* ankle-brachial pressure index <0.9 on one or both legs
* presence of leg artery disease with exertional leg symptoms (claudication)
* age 18-90 years

Exclusion Criteria:

* inability to provide written, informed consent
* medical conditions that make exercise testing unsafe (e.g. unstable angina)
* comorbidities that limit walking performance to a greater extent than claudication symptoms
* unable to complete the tests involved in the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with intermittent claudication recruited from hospital clinics
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2011-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Treadmill maximum walking distance | 2 weeks
EACH-Q walking questionnaire score | 2 weeks

SECONDARY OUTCOMES:
WIQ walking questionnaire score | 2 weeks
Self-reported maximum walking distance | 2 weeks
6-minute maximum walking distance | 2 weeks
GPS-measured maximum walking distance | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Garry A Tew, PhD, Principal Investigator — Sheffield Hallam University; Pierre Abraham, MD, PhD, Principal Investigator — University Hospital of Angers, France; Shah Nawaz, MD, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Sheffield Hallam University, Sheffield, South Yorkshire
  - Sheffield Vascular Institute, Sheffield, South Yorkshire

REFERENCES:
- [Derived] Tew G, Copeland R, Le Faucheur A, Gernigon M, Nawaz S, Abraham P. Feasibility and validity of self-reported walking capacity in patients with intermittent claudication. J Vasc Surg. 2013 May;57(5):1227-34. doi: 10.1016/j.jvs.2012.02.073. Epub 2013 Feb 4. PMID 23384490